CLINICAL TRIAL: NCT00788879
Title: Evaluation of a Media Campaign: Tu Salud Si Cuenta
Brief Title: Tu Salud Si Cuenta Media Campaign
Acronym: TSSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Belinda Reininger, Associate Professor, Health Promotion and Behavioral Sciences, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-05-0488; NIH NCMHD P20 MD000170-06
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Obesity; Diabetes
Keywords: Behavioral Journalism; Mexican-Americans; Obesity; Nutrition; Physical Activity; Border Health
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): This study arm is located in Brownsville, Texas. This community is exposed to the TSSC media messages as well as may be visited by the lay health workers and see the built environment changes
  Interventions: Behavioral: TSSC; Behavioral: TSSC Randomized Behavioral Intervention for weight loss
- 2 (No Intervention): The control group is located in Laredo. This community is not exposed to the TSSC messages nor does the campaign work to actively change the built environment or use lay health workers to share physical activity and nutrition information.

INTERVENTIONS:
Behavioral: TSSC — The intervention community is exposed to the media messages of the TSSC campaign. Residents of this community also receive the lay health worker visits as well as benefit from the positive built environment changes.
  Arms: 1
Behavioral: TSSC Randomized Behavioral Intervention for weight loss — We will enroll up to 200 weight-loss challenge participants to receive text messages on personal mobile phones throughout the challenge. Consent and enrollment in the trial will take place at registration for the weight-loss community challenge in the language of their choice. Recruited participants will be randomly assigned to a group after consenting to the study and the timing and content of text messages will vary according to group assignment (Groups A - D).
  Group A will receive weekly reminders for upcoming weigh-in events. Group B will receive the same weekly reminders but will also receive one-way messages every two weeks providing the participant motivational messages/topics and weight loss health tips. Group C will receive the same text messages as Group B but will also receive weekly prompts to self-monitor weight status. Group D will receive the same text messages as Group C plus daily prompts that will act as a guide for the participant to monitor behavior changes.
  Arms: 1

SUMMARY:
The Tu Salud, Si Cuenta (TSSC) media campaign uses behavioral journalism, community outreach and environmental changes to promote physical activity and nutritional changes among disadvantaged Mexican-Americans living along the U.S./Mexico border. This intervention posits that increased physical activity and increased fruit and vegetable consumption with smaller portion sizes will result in a decrease in obesity prevalence and diabetes incidence in this population.

DETAILED DESCRIPTION:
The TSSC campaign relies on behavioral journalism which includes the use of Spanish language, attractive and influential role models to illustrate healthy physical activity and nutritional habits through television, radio, and print media, to convey healthy physical activity and nutritional messages to the target population. This intervention method will be coupled with community outreach and environmental changes in the host community to further promote these changes. Community outreach includes the use of local, lay community workers to provide information and health screenings. Environmental changes focus on creating a positive built environment that promotes physical activity through well-lit streets, walking trails and safe recreational areas and healthy nutritional behaviors through increased access to markets and centers where affordable produce can be purchased and nutritional knowledge on healthy foods preparation and use can be disseminated.

As part of this intervention, a promoter-led community weight-loss challenge will be comprised of participants from the City of Brownsville's sixteen week weight-loss challenge. The location and site of the weigh-ins for this challenge occur at City Parks and Recreation facility on designated dates. Community members who select to participate in the city's weight loss challenge will be exposed to the Tu Salud Si Cuenta campaign. These individuals will have the same access to promoter-led exercise classes and nutrition education sessions, similar to CCHC participants. Recruited participants will also have the same access to information provided by promoters about health, physical activity and healthful food choices using motivational interviewing strategies. Participants of the weight-loss challenge are asked to weigh-in at least two times during the challenge and have their height, blood pressure and hip and waist circumference assessed.

We are proposing to evaluate the efficacy of this weight loss challenge more stringently and answer two important questions. The firs is what timing and types of support via text messages is appropriate for supporting weight loss in a community based weight loss challenge? The second question is what is the long term weight loss maintenance of participants in the 16 week weight loss challenge?

To answer the first question we will recruit and enroll Individuals who participate in the weight-loss challenge in a randomized behavioral intervention trial examining exposure to text messages and weight loss outcomes. Prior research has shown that making a change in behavior and weight loss can be dependent upon the type of messages provided to an individual (Rothman AJ, Salovey P, Antone C, et al, 1993; Patrick K, Raab F, Adams MA, 2009). We will test whether different content delivered via text messages impacts weight loss outcomes.

For this study, we will enroll up to 200 weight-loss challenge participants to receive text messages on their personal mobile phones throughout the 16 week challenge. Consent and enrollment in the trial will take place at registration for the weight-loss community challenge in the language of their choice. Recruited participants will be randomly assigned to a group after consenting to the study and the timing and content of text messages will vary according to group assignment (Groups A - D).

Group A will receive weekly reminders for upcoming weigh-in events. Group B will receive the same weekly reminders but will also receive one-way messages every two weeks providing the participant motivational messages/topics and weight loss health tips. Group C will receive the same text messages as Group B but will also receive weekly prompts to self-monitor weight status. The final group, Group D will receive the same text messages as Group C plus daily prompts that will act as a guide for the participant to monitor his or her behavior changes.

Participants will be asked to complete a short questionnaire about fruit and vegetable consumption, physical activity and social support for weight loss at the initial and final weigh in. (See attachment) We will also conduct a brief qualitative interview with 10 people per group about their opinions regarding the texting content and frequency. Finally, they will also consent for the research team to access their weight loss measures at initial and final weigh in and use in the research project to assess weight status changes. For those participants who do not attend final weigh in, the research team will contact the participant to obtain a final weight. At the time of enrollment into the behavioral intervention trial, participants will receive a $5 incentive. They will also receive an additional $10 incentive at the final weigh-in with their completed measures.

To answer the second research question of what is the long term weight loss maintenance of participants in the 16 week weight loss challenge we are proposing a follow-up feasibility study. We will enroll and consent Biggest Loser Challenge participants in a study that will follow them beyond the 16 week challenge one time at three months. At the registration of the weight-loss challenge participants will be consented in the language of their choice.

This study will enroll up to 150 consenting participants. Participants will have their height, weight, blood pressure and hip and waist circumference measures at initial, final weigh-in and 3 months post using the same protocols as all other Biggest Loser Challenge Participants. Weight will be taken using a calibrated Tanita scale and hip and waist circumference will be measured with a tape measure following protocols used in our CCHC (described below). Trained individual will take all measurements. A special number will be used to identify the participant in the study and only the investigator will know their name. These study participants however will also complete a short questionnaire about fruit and vegetable consumption, physical activity and social support for weight loss. (see attachment- this is the same instrument being used in the behavioral intervention trial examining text messaging)

For Biggest Loser Challenge participants who do not complete the final weigh-in measure but who have enrolled in this study, staff will contact the participants and schedule a time and location to obtain the final weigh in measures. The measures will need to be obtained within three weeks of the scheduled final weigh in challenge date. For the three month follow-up contact again we will contact the participant and schedule a time and location to obtain follow-up measures. Following all measurements (during the challenge and follow-up period), participants will have the opportunity to discuss their results with a community health worker trained to discuss these issues.

Individuals who complete the additional measures beyond the challenge period will receive incentives for their time associated with participating in the research study. Participants will receive an item valued at $5.00 for completing the three month post measurements.

ELIGIBILITY:
Inclusion Criteria:

* To be included in the evaluation survey study the participants must be living in Cameron park or Laredo TX at the time of the study, Hispanic men or women aged 20 - 75. The participants must speak Spanish.
* To be included in the observational study of physical activity the participants must be visiting the observational study site (park, exercise facility, walking trail) at the time of observation. No other criteria for inclusion exists for this study.
* To be included in the Randomized Behavioral Intervention, the participants must be participants in the weight-loss challenge and 18 years or older.

Exclusion Criteria:

* Participants who will be excluded from the evaluation survey study include those who are not Hispanic, not living in Cameron Park or Laredo TX, unable to speak Spanish and are either older than 55 or younger than 20.
* Participants excluded from the Randomized Behavioral Intervention are those younger than 18 and not participants of the weight loss challenge.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3100 (Actual)
Dates: Start 2003-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Physical Activity | baseline, yr. 3, post-intervention
Fruit and Vegetable Intake | baseline, yr. 3, post-intervention

SECONDARY OUTCOMES:
Waist circumference | baseline, yr. 3, post-intervention
Hip circumference | baseline, yr. 3, post-intervention
Confirmed Awareness: Confirmation of recognition of messages | baseline, third year, post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Belinda M Reininger, DrPH, Principal Investigator — University of Texas Houston Health Science Center; Kevin Hwang, MD, Principal Investigator — University of Texas Medical School
Locations (1):
- University of Texas Houston Health Science Center, Brownsville Regional Campus, Brownsville, Texas, United States

REFERENCES:
- [Result] Reininger BM, Barroso CS, Mitchell-Bennett L, Cantu E, Fernandez ME, Gonzalez DA, Chavez M, Freeberg D, McAlister A. Process evaluation and participatory methods in an obesity-prevention media campaign for Mexican Americans. Health Promot Pract. 2010 May;11(3):347-57. doi: 10.1177/1524839908321486. Epub 2009 Jan 8. PMID 19131541
- [Derived] Heredia NI, Lee M, Reininger BM. Exposure to a community-wide campaign is associated with physical activity and sedentary behavior among Hispanic adults on the Texas-Mexico border. BMC Public Health. 2017 Nov 16;17(1):883. doi: 10.1186/s12889-017-4893-4. PMID 29145821